CLINICAL TRIAL: NCT05052515
Title: The Effects of Natural Extract With Dihydromiricetin on MASLD Patients
Brief Title: The Effects of Dihydromiricetin on MASLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Papatheodoridis, Professor in Medicine & Gastroenterology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 436/14-06-21
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: NAFLD
Keywords: dihydromiricetin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ascorbic Acid; Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Oral treatment Two capsules twice daily for one year
  Interventions: Other: Placebo
- Nutritional Supplementation (Experimental): Oral treatment Two capsules twice daily for one year
  Interventions: Dietary Supplement: Dihydromiricetin, Vitamin C, E and Choline

INTERVENTIONS:
Dietary Supplement: Dihydromiricetin, Vitamin C, E and Choline — Patients with MASLD will be randomly allocated to receive capsules with Dihydromiricetin, Vitamin C, E and Choline
  Arms: Nutritional Supplementation
Other: Placebo — Patients with MASLD will be randomly allocated to receive placebo capsules
  Arms: Placebo

SUMMARY:
The global wave of obesity has affected dramatically the incidence of non-alcoholic fatty liver disease (NAFLD) making it the leading cause of liver disease in the western world. NAFLD is considered the hepatic manifestation of metabolic syndrome and is strongly associated with type II diabetes, sleep apnea and cardiovascular disease. Although cardiovascular disease is the leading cause of death in patients with NAFLD, a subset of patients who meet the histological criteria for steatohepatitis have the highest risk for liver-related morbidity and mortality.

Reviewing literature, it appears that several pathophysiologic mechanisms related to metabolism, inflammation and fibrosis are deregulated in NAFLD, whereas dihydromiricetin natural extracts have been suggested to exhibit antioxidant activity. In contrast to Vitamin E, which has been studied as an agent for non-diabetic patients with NAFLD, epidemiological and/or clinical data for the use of dihydromiricetin natural extracts or their combination in NAFLD are limited.

DETAILED DESCRIPTION:
The study will be randomized, placebo-controlled and double-blinded in order to avoid systemic errors, such as selection bias and the placebo effect. Patients will be randomly assigned to one of two groups: A) capsules with dihydromiricetin, vitamins C/E and choline (two capsules per day) and B) placebo (identical capsules). The duration of the intervention will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Alanine aminotransferase (ALT) higher than the upper limit of normal with or without elevated γ-glutamyl transpeptidase (γGT)
* Hepatic steatosis-indicating findings on ultrasound and / or liver biopsy
* BMI 20-45 Kg/m2

Exclusion Criteria:

* Alcohol consumption > 210 or > 140 grams per week for men or women, respectively
* Use of a potentially hepatotoxic drug
* Detection of hepatitis B virus (HBsAg) surface antigen or Hepatitis C virus antibodies (anti-HCV) or HIV antibodies
* The coexistence of α systemic disease with potentially hepatic involvement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
ALT change | 12 months.
  ALT normalization or reduction of ALT >50% compared to baseline

SECONDARY OUTCOMES:
ALT and GGT changes | 6 and 12 months
  Normalization of both ALT and GGT
Liver stiffness change | 12 months
  Change of liver stiffness at liver elastography by >1 kPa

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Papatheodoridis, MD PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- General Hospital of Athens "Laiko", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No